CLINICAL TRIAL: NCT05024253
Title: Does Perioperative Use of Tranexamic (TXA) in Bone Tumor Surgery Reduce Blood Loss and Transfusion Requirements? A Double-blinded Randomized Controlled Trial
Brief Title: Perioperative Use of Tranexamic (TXA) in Bone Tumor Surgery Will Change in Blood Loss and Transfusion Requirements.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCHE-BoneT003
Record Dates: First submitted 2021-08-17; First posted 2021-08-27 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2022-10

CONDITIONS: Ewing Sarcoma of Bone; Osteosarcoma
Keywords: tranexamic acid
MeSH Terms: conditions — Osteosarcoma | interventions — Tranexamic Acid; Sodium Chloride; Fluoridation

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, double-blinded clinical trial will be done on all included case. They will be divided into two groups based randomly using Block Stratified Randomized Software program, after obtaining informed consent from eligible patient or his caregiver into two Arms:
  Arm A: patient is not receiving TXA but instead receiving a placebo (saline injection) Arm B: patient is receiving TXA which is colorless solution.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The PI, primary surgeon, anesthesiologist, patient, all assisting surgeons and anesthesiologist as well operating and circulating nurse will be blinded to the study arm to which patient belongs to. Only clinical trial unit and pharmacist will be unblinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patient is receiving Tranexemic acid (TXA ) (Experimental): Loading dose: Prior to surgical incision, and according to allocated arm, pharmacist will prepare TXA injection at a dose of 10mg/kg diluted in 50ml normal saline (maximum concentration 100mg/ml).
  Maintenance dose: Throughout surgery, continuous infusion at a dose of 5mg/kg/hour will be given until wound closure.
  Interventions: Drug: Tranexamic acid injection
- standard treatment (saline) (Placebo Comparator): Loading dose: Prior to surgical incision, and according to allocated arm, pharmacist will prepare 50 ml of 0.9% saline or TXA at a dose of 10mg/kg diluted in 50ml normal saline (maximum concentration 100mg/ml).
  Maintenance dose: Throughout surgery, continuous infusion of saline will be given until wound closure.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Tranexamic acid injection — . TXA, a lysine analogue, reversibly binds to the plasminogen lysine receptors and thereby blocks plasminogen from binding to fibrin (tPA can only activate fibrin-bound plasminogen and produce plasmin responsible for cleaving fibrin molecule and dissolving the blood clot)
  Other Names: Cyklokapron®
  Arms: patient is receiving Tranexemic acid (TXA )
Other: Saline — mixture of sodium chloride (salt) and water in solution with 0.90% w/v of NaCl
  Other Names: Salt water
  Arms: standard treatment (saline)

SUMMARY:
The purpose of this trial is to investigate whether previously reported benefit of Tranexamic acid in pediatric orthopedic surgeries could be recapitulated in bone tumor surgeries or not through a double blinded randomized controlled trial done in children cancer hospital 57357.

DETAILED DESCRIPTION:
Resection of bone tumors is commonly associated with considerable intra and post-operative blood loss due to extensive soft tissue dissection, multiple bone osteotomies, prolonged operative time. The intraoperative use of limb tourniquet to reduce bleeding may not be applicable in all situations e.g. arm, thigh and pelvic surgeries. The use of cell savers for auto transplantation of blood is not preferred in cancer surgeries. Antifibrinolytic drug are currently used to reduce perioperative blood loss in a variety of orthopedic surgeries. Currently, the most common agents used are EACA and TXA. A third agent, aprotinin, was withdrawn from the market in 2007 owing to safety concerns noted in several studies, suggesting an increased risk of death and renal dysfunction in patients undergoing cardiac surgery. Slow to adopt in obstetric population, TXA became popular for patients with hereditary bleeding disorders for whom menorrhagia, frequent spontaneous nose bleeds, or dental procedures could be life threatening. With strong record as an effective and safe medicine, TXA has earned its place on the World Health Organization List of Essential Medicines as an important drug needed in every health system. More recently, its use has expanded to treat or prevent excessive blood loss from trauma and major surgery, including cardiac, orthopedic, and hepatic procedures. TXA, a lysine analogue, reversibly binds to the plasminogen lysine receptors and thereby blocks plasminogen from binding to fibrin (tPA can only activate fibrin-bound plasminogen and produce plasmin responsible for cleaving fibrin molecule and dissolving the blood clot) TXA has been extensively studied in joint replacement surgeries specifically total knee replacement, scoliosis surgery, and in trauma surgeries. The question of efficacy of TXA in these surgeries was addressed in multiple prospective randomized studies and subsequent meta-analysis. Main concern regarding increased risk of DVT was negated in several of these studies. The American Academy of Orthopedic Surgeons provides a strong recommendation for the use of any administration of TXA for joint arthroplasty and states that it does not seem to increase the risk of thromboembolic or myocardial complications. Junlong Zhong et al. in 2019 published a systematic review and meta-analyses on 2500 pediatric patients undergoing corrective surgery for idiopathic scoliosis. They concluded that TXA was effective in reducing surgical time, intraoperative blood loss and blood transfusion without increasing complications. Levack et al. Published in 2020 a randomized controlled trial on role of TXA in reducing blood loss and transfusion in pediatric patients undergoing a periacetabular osteotomy. They concluded that TXA reduced blood loss by 293ml and reduced frequency of allogenic transfusions by 73%.

The purpose of this trial is to investigate whether previously reported benefit of Tranexamic acid in pediatric orthopedic surgeries could be recapitulated in bone tumor surgeries or not through a double blinded randomized controlled trial done in children cancer hospital 57357.

ELIGIBILITY:
Inclusion Criteria:

1. Malignant bone tumor of the femur and finished neoadjuvant chemotherapy
2. Candidate for resection and reconstruction by prosthesis. 3- Age 4-18 years.

Exclusion Criteria:

1. Anatomic location other than femur de
2. Reconstruction other than prosthesis
3. Allergy to TXA
4. Previous history of DVT
5. Previous history of renal dysfunction
6. Congenital or acquired coagulopathy.
7. Congenital or acquired cardiomyopathy.
8. Previous history of convulsions.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss will be changed by by Tranexamic acid when compared with saline or Not. | during surgery
  will be calculated based on measurement of number and weights of blood-soaked surgical swabs. As well as measurement of total volume of blood collected in suction container, after subtracting volume of saline used for washing wound.
postoperative blood loss will be changed by Tranexamic acid when compared with saline or Not. | after surgery , approximately 1-4 days
  will be calculated based on measurement of number and weights of blood-soaked surgical swabs. As well as measurement of total volume of blood collected in suction container, after subtracting volume of saline used for washing wound.

SECONDARY OUTCOMES:
blood transfusion will be changed by Tranexamic acid when compared with saline or Not. | during surgery and approximately 1-7 days
  Calculation of blood volume to be transfused (no of units in mls) = (Estimated blood volume ×(target HCT -actual HCT))/HCT of one unit of packed RBCs

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M ELGHONEIMY, MD, Principal Investigator — 57357 children cancer hospital
Locations (1):
- Children's Cancer Hospital Egypt 57357 Cairo, Egypt, Cairo, Egypt

REFERENCES:
- [Background] Levack AE, McLawhorn AS, Dodwell E, DelPizzo K, Nguyen J, Sink E. Intravenous tranexamic acid reduces blood loss and transfusion requirements after periacetabular osteotomy. Bone Joint J. 2020 Sep;102-B(9):1151-1157. doi: 10.1302/0301-620X.102B9.BJJ-2019-1777.R1. PMID 32862676
- [Background] Dadure C, Sauter M, Bringuier S, Bigorre M, Raux O, Rochette A, Canaud N, Capdevila X. Intraoperative tranexamic acid reduces blood transfusion in children undergoing craniosynostosis surgery: a randomized double-blind study. Anesthesiology. 2011 Apr;114(4):856-61. doi: 10.1097/ALN.0b013e318210f9e3. PMID 21358317
- [Background] Carabini LM, Moreland NC, Vealey RJ, Bebawy JF, Koski TR, Koht A, Gupta DK, Avram MJ; Northwestern High Risk Spine Group. A Randomized Controlled Trial of Low-Dose Tranexamic Acid versus Placebo to Reduce Red Blood Cell Transfusion During Complex Multilevel Spine Fusion Surgery. World Neurosurg. 2018 Feb;110:e572-e579. doi: 10.1016/j.wneu.2017.11.070. Epub 2017 Nov 22. PMID 29175569
- [Background] Johnson DJ, Johnson CC, Goobie SM, Nami N, Wetzler JA, Sponseller PD, Frank SM. High-dose Versus Low-dose Tranexamic Acid to Reduce Transfusion Requirements in Pediatric Scoliosis Surgery. J Pediatr Orthop. 2017 Dec;37(8):e552-e557. doi: 10.1097/BPO.0000000000000820. PMID 29120963